CLINICAL TRIAL: NCT03910829
Title: Effects of Motor Imagery and Action Observation Training on Neck Reposition Sense in Patients With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6
Record Dates: First submitted 2019-04-02; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Chronic Pain
Keywords: Motor Imagery; Action observation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Action Observation (Experimental): This group receives an action observation training through the visualization of a video of cervical movements.
  Interventions: Behavioral: Action Observation
- Motor Imagery (Experimental): This group receives an motor imagery through the imagery process of cervical movements.
  Interventions: Behavioral: Motor Imagery
- Placebo Group (Placebo Comparator): This group receives a placebo action observation training through the visualization of a video of a documentary video
  Interventions: Behavioral: Placebo Action Observation

INTERVENTIONS:
Behavioral: Action Observation — Action observation training
  Arms: Action Observation
Behavioral: Motor Imagery — Motor imagery protocol
  Arms: Motor Imagery
Behavioral: Placebo Action Observation — Placebo Action Observation
  Arms: Placebo Group

SUMMARY:
This study evaluates the influence of motor imagery or action observation training on joint position error in patients with chronic neck pain. This variable is a measure of proprioception and cervical motor control. A group of patients will receive an action observation training of neck movements, another will receive a protocol of motor imagery of the same movements and the last group will be a placebo group, through the viewing of a documentary video.

DETAILED DESCRIPTION:
Motor imagery is defined as a dynamic mental process of an action, without its real motor execution. Action observation training consists of watching an action performed by someone else. Both motor imagery and action observation have been shown to produce a neurophysiological activation of the brain areas related to the planning and execution of voluntary movement in a manner that resembles how the action is performed in reality.

Both motor imagery and action observation are interventions that can generate adaptive neuroplastic changes on a cortical level, leading to a decrease in chronic pain. These rehabilitation techniques are used in pain treatment and impaired movement injuries that could be due to a nervous system alteration.

The effectiveness of motor imagery is controversial; several studies have presented unfavorable outcomes from this technique. Some variables, such as the duration of the sessions, the time employed the type of motor task or the number of sessions can influence the outcomes of these studies. Thus, it is necessary to clarify the controversial aspects of motor imagery, which lead us to perform this study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 65 years
* Medical diagnosis of NSCNP with more than 6 months of evolution of neck pain

Exclusion Criteria:

* Patients with rheumatic diseases, cervical hernia, cervical whiplash syndrome, neck surgeries o a history of arthrodesis
* Systemic diseases
* Vision, hearing or vestibular problems
* Severe trauma or a traffic accident that had an impact on the cervical area.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-15 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Joint Position Error (JPE) | Change from baseline and immediately post-intervention
  JPE will be assessed with Motion Guidance Clinic Kit. This device consisted of adjustable straps and a fastening support for a laser beam. Patients were asked to sit in a comfortable position at a 90-cm distance from the bullseye with the device correctly placed. With eyes closed, they were asked to point to the neutral position of the head and memorize. This point was recorded as a reference for each patient. The patient subsequently performed a maximal movement of cervical flexion and then attempted to find the initial reference position with a maximum of precision without speed instruction. The point on which the light beam stopped indicated the global error measured in centimeters (cm) in relation to the center of the target recorded previously. The same protocol was used for the extension, right and left rotation movements. Ten trials were performed with head repositioning after each movement, and the mean measure was recorded.

SECONDARY OUTCOMES:
Visual and Kinesthetic Motor Imagery Ability | Immediately before the intervention
  Visual and Kinesthetic Motor Imagery Ability will be measured with Movement Imagery Questionnaire-Revised (MIQ-R). MIQ-R has four movements repeated in two subscales, a visual and a kinesthetic one. Additionally, a score between 1 and 7 is assigned, with 1 representing difficulty in picturing the motor image or difficulty in feeling the movement previously made, and 7 representing the maximum ease. The internal consistencies of the MIQ-R have been consistently adequate with Cronbach's α coefficients ranging above 0.84 for the total scale, 0.80 for de visual subscale and 0.84 for the kinesthetic subscale (Campos & González, 2010).
Mental Chronometry | Immediately before the intervention
  Mental chronometry evaluation was also used to measure the subject's motor imagery
The degree of physical activity | Immediately before the intervention
  The degree of physical activity was objectified through the IPAQ questionnaire, which allows the subjects to be divided into three groups according to their level of activity, which can be high, moderate, and low or inactive (Roman-Viñas et al., 2010). This questionnaire has shown an acceptable validity to measure total physical activity. Therefore, the psychometric properties of the questionnaire were accepted for use in studies that required the measurement of physical activity.
Laterality task | Immediately before the intervention
  With the task of recognition of the neck's laterality, two aspects will be evaluated: first, the precision (percentage of correct answers) of the discrimination of the laterality which is the capacity to recognize if a part of the body belongs to the right or left and second, the response time that the participants use in the task of discrimination or cognitive judgment. The app designed and developed by the NOI group will be used.
Pain catastrophizing | Immediately before the intervention
  The Spanish version of the pain catastrophizing scale (PCS) assesses the degree of pain catastrophizing. The PCS has 13 items and a 3-factor structure of rumination, magnification, and helplessness.
Kinesiophobia | Immediately before the intervention
  Fear of movement or kinesiophobia will be quantified with the Spanish version of the Kinesiophobia Tampa Scale (TSK-11). This instrument demonstrates reliability and validity in patients with chronic pain, being shorter than the original scale. The total score ranges from 11 to 44 points, with the highest scores indicating greater fear of a new injury due to movement

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain